CLINICAL TRIAL: NCT02509221
Title: Effect of Duration of Exposure of Anesthesia With Sevoflurane on Emergence Delirium
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Joseph Resti, MD, State University of New York - Upstate Medical University
Other Study IDs: 714457
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Delirium on Emergence
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Less than 30 minutes
- 30-60 minutes
- More than 60 minutes

SUMMARY:
Emergence delirium which is a phenomenon seen commonly in preschool kids anesthetized with Sevoflurane. Restless recovery from anesthesia may not only cause injury to the child or to the surgical site, but may also lead to the accidental removal of surgical dressings, IV catheters, and drains. is one of the The purpose of the study is to find whether duration of exposure to Sevoflurane has any effect on the incidence of Emergence Delirium.

ELIGIBILITY:
Inclusion Criteria:

* age between 1-6 years of age
* receiving general anesthesia for non-surgical procedure

Exclusion Criteria:

* history of emergence delirium
* severe CNS disease

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients between 1-6 years old receiving anesthesia for non-surgical reasons
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Incidence of emergence delirium | 30 mintes after anesthesia
  using the PAED scale
Severity of emergence delirium | 30 minutes after anesthesia
  using the PAED scale

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Syracuse, New York, United States